CLINICAL TRIAL: NCT06546384
Title: Effect of Glucagon-like Peptide-1 Receptor Agonists (GLP-1 RA) on Alcohol Consumption, Metabolism and Liver Parameters in Patients With Obesity and Fatty Liver Disease
Brief Title: GLP-1 RA on Alcohol Consumption, Metabolism and Liver Parameters in Patients With Obesity and Fatty Liver Disease
Acronym: GLP-1 RA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01715
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Adiposity; Fatty Liver; Alcohol Use Disorder
Keywords: GLP-1; Semaglutide
MeSH Terms: conditions — Obesity; Fatty Liver; Alcoholism | interventions — semaglutide; Exercise

STUDY DESIGN:
Intervention Model Description: This is an exploratory, monocentric, randomized controlled clinical trial
Masking Description: No blinding procedures in place
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide Arm (Experimental): Patients assigned to this arm will be treated with semaglutide and standard of care for weight reduction (nutritional and exercise recommendations) for 16 weeks.
  Interventions: Drug: Semaglutide; Behavioral: Weight reduction recommendations (nutritional and exercise)
- Control Arm (Active Comparator): Patients assigned to this arm will be treated with standard of care for weight reduction (nutritional and exercise recommendations) for 16 weeks.
  Interventions: Behavioral: Weight reduction recommendations (nutritional and exercise)

INTERVENTIONS:
Drug: Semaglutide — Treatment with semaglutide, following standard clinical practice as per below schedule:
  Week 1-4: Injected dose of 0,25 mg i.d. Week 5-8: Injected dose of 0,5 mg i.d. Week 9-12: Injected dose of 1,0 mg i.d. Week 13-16: Injected dose of 1,7 mg i.d. After week 16: Injected dose of 2,4 mg i.d.
  Arms: Semaglutide Arm
Behavioral: Weight reduction recommendations (nutritional and exercise) — Participants will receive nutritional and exercise recommendations and 2 telephone consultations

SUMMARY:
There is evidence that alcoholic beverage consumption significantly interacts with food energy intake. Furthermore, there is accumulating evidence showing independent, combined, and modifying effects of alcohol and metabolic factors on the onset and progression of chronic liver disease. Preclinical and clinical data have showed that GLP-1 RA can decrease alcohol consumption, particularly in obese patients. Moreover there is evidence that semaglutide can improve the liver sinusoidal milieu in pre-clinical models of cirrhosis.

In this study, the investigators aim to assess if patients treated with semaglutide and receiving counselling will achieve a significantly higher alcohol abstinence compared to patients only receiving counselling.

DETAILED DESCRIPTION:
In Switzerland, approximately 20% of the population is consuming more alcohol than recommended by the WHO. There is evidence that alcoholic beverage consumption significantly interacts with food energy intake. Although several studies have investigated the role of alcohol in obesity, there is still a lack of knowledge about specific roles of different types of alcoholic beverages and on the effect of consumption patterns in patients with metabolic syndrome and obesity. Nevertheless, there is accumulating evidence showing independent, combined, and modifying effects of alcohol and metabolic factors on the onset and progression of chronic liver disease.

Glucagon-like peptide-1 (GLP-1)-based therapy for type 2 diabetes was introduced in 2006. GLP-1 is an incretin hormone, which is secreted from endocrine L cells of the small intestine in response to nutrients in the gut lumen. Exendin-4 binds to the GLP-1R with high affinity and acts as a receptor agonist, thus referred to as GLP-1 receptor agonists (GLP-1 RA). To date the GLP-1 RA: dulaglutide, semaglutide, liraglutide, lixisenatide and exenatide are approved for the treatment of diabetes mellitus type II in Switzerland. Since 2020, the GLP-1 RA semaglutide is also approved for the treatment of obesity in Switzerland. GLP-1 RA have a well-established effect on the food reward system which is regulated by key mesolimbic brain regions, the ventral tegmental area (VTA) and nucleus accumbens (NAc)11. Interestingly, these regions are also involved in the rewarding effects of drugs of abuse and alcohol. A link between alcohol intake and GLP-1 has been demonstrated in several preclinical studies and may play an important role in the development of addiction. The findings are consistent with the hypothesis that systemic administration of GLP-1 RA can influence the mesolimbic dopamine system and reward-seeking behaviours associated with alcohol use disorder (AUD). Furthermore, preclinical data has shown that GLP-1 RA, namely, liraglutide significantly improved liver microvascular function and exhibited anti-fibrotic effects of confirmed in human liver tissue.

In metabolic fatty liver disease, GLP-1 RA have a significant effect on reducing steatosis and inflammation. Obesity is one of the main risk factors for fatty liver disease, particularly central adiposity, and one of the leading drivers for liver disease progression, independent of the cause of liver disease. In a Swiss referral liver centre, 75% of patients with advanced cirrhosis have either alcohol, metabolic or combined factors (25%) as the cause for liver disease. Therapeutic strategies approaching both aetiologies are thus urgently needed.

The investigators aim to investigate in this study, whether there is a significant beneficial effect of GLP-1 RA, specifically semaglutide, on alcohol consumption, specifically in obese patients. Furthermore, the investigators aim to systematically assess drinking patterns and alcohol beverage consumption in patients with obesity assessed with the innovative direct alcohol biomarker phosphatidylethanol (PEth)24 that overcomes the problems of low reliability of medical history, standard questionnaires and previous tests in assessing recent alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m² OR BMI ≥ 28 kg/m² in the case of weight-related co-morbidities (pre-diabetes or type 2 diabetes mellitus, hypertension, dyslipidemia).
* Fatty liver disease (steatosis on ultrasound and/or CAP value on FS > 238 dB/m)
* Age 18 - 80 years
* Alcohol Use Disorder Identification Test-C Score >4 (AUDIT-C) Score ≥4 for women and ≥5 for men (as measured from AUDIT-questionnaire distributed in visit 1)
* Sufficient skills for German or French language (written and spoken)
* Signed informed consent

Exclusion Criteria:

* Active illicit substance use
* AUDIT-score < 5 (males)/ 4 (females) (as measured from AUDIT-questionnaire distributed in visit 1)
* Current treatment with drugs against alcohol dependence (disulfiram, acamprosate, naltrexone, baclofen and nalmefene)
* Any known contraindication to semaglutide
* Presence or history of a hepatic or extrahepatic malignancy from the previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving total alcohol abstinence (measured by negative PEth test) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Percentage of patients achieving total alcohol abstinence from baseline to follow-up after 16 weeks of treatment, measured by negative PEth test, in patients treated with semaglutide vs control.

SECONDARY OUTCOMES:
Proportion of patients achieving total alcohol abstinence (measured by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Percentage of patients achieving total alcohol abstinence from baseline to follow-up after 16 weeks of treatment, measured by TFLB method, in patients treated with semaglutide vs control.
Proportion of patients maintaining total alcohol abstinence (measured by negative EtG) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Percentage of patients maintaining total alcohol abstinence from baseline to follow-up after 16 weeks of treatment, measured by negative EtG in patients treated semaglutide vs. control
Change of alcohol abstinent days (cumulative abstinent days, by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Assessment of change in percentage of alcohol abstinent days after treatment compared to before treatment with semaglutide vs. control (measured by TFLB method)
Change of heavy drinking days (by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Assessment of change in percentage of heavy drinking days after treatment compared to before treatment with semaglutide vs. control (measured by TFLB method)
Change of total number of drinks per week (by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Assessment of change in percentage of total number of drinks per week after treatment compared to weeks before treatment with semaglutide vs. control (measured by TFLB method)
Pre and post treatment comparison of total abstinence (PEth test) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Change from baseline in number of patients with total alcohol abstinence as assessed by PEth test.
Pre and post treatment comparison of total abstinence (assessed by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Change from baseline in number of patients with total alcohol abstinence as assessed by TFLB method.
Pre and post treatment comparison of total abstinence (measured by negative EtG) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Change from baseline in number of patients with total alcohol abstinence measured by negative EtG.
Pre and post treatment comparison of cumulative abstinent days (by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Change from baseline in number of cumulative abstinent days per patient (measured by TFLB method).
Pre and post treatment comparison of drinking days (by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Change from baseline in number of drinking days per patient (measured by TFLB method).
Pre and post treatment comparison of number of drinks per week (by TFLB method) | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Change from baseline in number of drinks per week per patient (measured by TFLB method).
Effects of semaglutide on reward and relief drinking behavior | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Assessments of effects of semaglutide on reward and relief drinking behavior (assessed with the Alcohol Expectancy Questionnaire, both study arms).
Percentage reduction in transient liver elastography levels assessed by Fibroscan | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Percentage reduction in transient liver elastography levels by vibration controlled transient elastography (Fibroscan) from baseline until after 16 weeks of therapy (both study arms).
Percentage reduction in transient liver elastography levels assessed by FIB-4 score | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Percentage reduction in transient liver elastography levels by FIB-4 score (fibrosis assessment including age, AST, ALT and platelet count) from baseline until after 16 weeks of therapy (both study arms).
Percentage reduction in metabolic markers | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Percentage reduction in metabolic markers (both study arms): body weight, BMI, fasting glucose, homeostatic model assessment of insulin resistance (HOMA-IR), HbA1c levels from baseline until 16 weeks after therapy
Safety profile of semaglutide in described population | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Number and description of SAE's concerning semaglutide in described population (semaglutide arm only).
Effect of GLP-1 RA therapy on TMA/TMAO pathway | From inclusion date (baseline) until end of the study, total duration 16 weeks per patient
  Statistically significant % reduction of TMAO levels (measured by blood test at baseline and after 16 weeks of therapy, semaglutide arm only).

CONTACTS AND LOCATIONS:
Overall Officials: Susana Gomes Rodrigues, MD, Principal Investigator — University Hospital Bern (Inselspital), Hepatology
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No